CLINICAL TRIAL: NCT03587194
Title: A Single Center Study to Evaluate the Effectiveness and Safety of Add on Enstilar® in Patients Using OTEZLA® for Moderate to Severe Plaque Psoriasis
Brief Title: Evaluation of Add on Enstilar in Patients Using Otezla for Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP-CL-PSOR-PI-13156
Record Dates: First submitted 2018-07-02; First posted 2018-07-16 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Otezla Enstilar (Experimental): Otezla 30mg BID Enstilar QD
  Interventions: Drug: Otezla

INTERVENTIONS:
Drug: Otezla — Otezla 30mg BID

SUMMARY:
Add-on Enstilar to Otezla therapy.

DETAILED DESCRIPTION:
50 adult patients with moderate to severe plaque psoriasis will be given OTEZLA® for 16 weeks with add-on Enstilar.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult ≥ 18 years of age;
2. Diagnosis of chronic plaque-type psoriasis
3. Moderate to severe plaque type psoriasis as defined at baseline by:

   * PGA score of 3 or greater
   * BSA affected by plaque-type psoriasis of 10% or greater
   * PASI ≥ 12
4. Able and willing to give written informed consent prior to performance of any study-related procedures
5. Must be in general good health (except for disease under study) as judged by the Investigator, based on medical history, physical examination, clinical laboratories, and urinalysis. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).

Exclusion Criteria:

1. Other than psoriasis, any clinically significant (as determined by the investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is uncontrolled.
2. Forms of psoriasis other than chronic plaque-type (e.g., Pustular erythrodermic and/or guttate psoriasis) or drug induced psoriasis
3. Subjects who previously used any biologic agent for psoriasis.
4. Use of oral systemic medications for the treatment of psoriasis within 4 weeks (includes, but not limited to, oral corticosteroids, methotrexate, acitretin and cyclosporine).
5. Patient used topical therapies to treat psoriasis on the hands and/or feet within 2 weeks of the Baseline Visit (includes, but not limited to, topical corticosteroids, vitamin D analogs, or retinoids).
6. Patient received UVB phototherapy within 2 weeks of Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Bagel, Principal Investigator — dreamacres1@aol.com
Locations (1):
- Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Otezla Enstilar: Otezla: Otezla 30mg BID Enstilar QD
Period: Overall Study
Arm/Group | Otezla Enstilar
Started | 50
Completed | 23
Not Completed | 27

BASELINE CHARACTERISTICS:
Arm/Group | Otezla Enstilar
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 48 [21 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area Severity Index 75 at Week 12
Description: Patients who achieve Psoriasis Area Severity Index 75 at week 12. PASI scores range 0-72 (maximal disease)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Otezla Enstilar
Number analyzed (Participants) | 31
Participants | 29

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Otezla Enstilar
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 7/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Otezla Enstilar (N=31)
mastoiditis (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Otezla Enstilar (N=31)
diarrhea (Gastrointestinal disorders) | 5 (5)
nausea (Gastrointestinal disorders) | 4 (4)
folliculitis (Skin and subcutaneous tissue disorders) | 2 (2)
leg pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Verrucous acanthoma (Skin and subcutaneous tissue disorders) | 1 (2)
vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT03587194/Prot_SAP_000.pdf